CLINICAL TRIAL: NCT04527354
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Pilot Study of Treamid Efficacy and Safety in the Rehabilitation of Patients After COVID-19 Pneumonia
Brief Title: Pilot Study to Assess Efficacy and Safety of Treamid in the Rehabilitation of Patients After COVID-19 Pneumonia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PHARMENTERPRISES LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COVID-TRE-03
Record Dates: First submitted 2020-08-24; First posted 2020-08-26 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: SARS-CoV-2 Infection; Fibrosis Lung
Keywords: COVID-19; Coronavirus; Rehabilitation
MeSH Terms: conditions — COVID-19; Pulmonary Fibrosis; Coronavirus Infections | interventions — N,N'-bis(2-(1H-imidazol-2-yl)ethyl)pentanediamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A blind will be performed by using Placebo equivalent to Treamid tablets without active substance and the corresponding labeling of the study drug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treamid 50 mg (Experimental): 1 tablet of Treamid 50 mg once a day during 4 weeks of treatment period.
  Interventions: Drug: Treamid
- Placebo (Placebo Comparator): 1 tablet of Placebo once a day during 4 weeks of treatment period
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treamid — Participants will receive Treamid 50 mg once a day during 4 weeks
  Arms: Treamid 50 mg
Drug: Placebo — Participants will receive Placebo once a day during 4 weeks
  Arms: Placebo

SUMMARY:
The innovative drug Treamid is planned for use in the rehabilitation of patients after COVID-19 pneumonia in a pilot, multicenter, randomized, double-blind, placebo-controlled Phase II clinical study to assess the efficacy and safety of Treamid, tablets, 50 mg in patients with fibrotic changes in the lungs after COVID-19 pneumonia during a 28-day treatment.

The primary objective of the study is to demonstrate the efficacy of Treamid tablet, 50 mg in change in forced vital capacity (FVC) and/or diffusing capacity of lung for carbon monoxide (DLCO) at Week 4.

The secondary objective of the study is to evaluate the safety of Treamid tablet, 50 mg and pharmacokinetics (PK).

DETAILED DESCRIPTION:
12-15 Russian centers are planned for participation in this pilot study. The study consists of three periods: screening (2 weeks), treatment period (4 weeks) and follow-up period (2 weeks after completion of treatment with Treamid / Placebo). The duration of participation in the study for each patient is no more than 8 weeks.

60 patients with fibrotic changes in the lungs after COVID-19 pneumonia are planned to be randomized. All patients will undergo a qualitative determination of coronavirus severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) by polymerase chain reaction (PCR). Patients will be evaluated using the Modified British Medical Research Council (mMRC) Dyspnea Scale, chest computed tomography (CT), spirometry and body plethysmography with determination of DLCO. This examination should be conducted as close as possible to the expected randomization date (no earlier than 5 days before). All eligible patients will be randomized into 2 groups in a 1:1 ratio: Treamid 50 mg daily (30 patients); Placebo (30 patients).

During the treatment period (4 weeks), patients will receive 1 tablet Treamid / Placebo once a day. Patients will be advised to continue the standard program of medical rehabilitation under day inpatient or outpatient conditions (stage 3 according to the Interim Guidelines for Medical Rehabilitation after New Coronavirus Infection (COVID-19), 2020.

Patients will visit the study center once a week. At the Week 1, Week 2 and Week 3 visits, Adverse events (AEs) and concomitant therapy, investigational drug registration, body weight, vital signs and Oxygen saturation (SpO2) scores, mMRC dyspnea score and spirometry will be recorded.

During the Week 2 visit, physical examination, electrocardiography (ECG), complete blood count (CBC) and biochemical blood test, PK study, common urine analysis, bodyplethysmography with DLCO will also be conducted. Patients will complete the KBILD questionnaire. Also, the patients will undergo a 6-minute walk test to measure the distance the patient walks for 6 minutes and evaluate using the Borg Scale. At the Week 4 visit (the end of the therapy), registration of AEs and concomitant therapy, physical examination, measurement of height, body weight, vital signs and SpO2, ECG, CBC and biochemical blood tests, PK study and common urine analysis will be conducted. Patients will be evaluated using the mMRC Dyspnea Scale, chest CT, spirometry and body plethysmography with determination of DLCO. Patients will complete the King's Brief Interstitial Lung Disease Questionnaire (KBILD) followed by a 6-minute walk test to measure the distance the patient walks for 6 minutes and evaluate using the Borg Scale.

Patient follow-up will continue for another 2 weeks. At the Week 6 visit, registration of AEs and concomitant therapy, physical examination, measurement of height, body weight, vital signs and SpO2, ECG, mMRC dyspnea score, CBC and biochemical blood tests, and common urine analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Signed patient explanation sheet and informed consent for participation in the study.
2. Men and women at the age from 18 through 75 years old.
3. Fibrous changes in the lungs after COVID-19 pneumonia:

   1. COVID-19 diagnosis in the past medical history confirmed by positive qualitative analysis of SARS-CoV-2 RNA by PCR method;
   2. The first symptoms of COVID-19 appear no earlier than 2 months before the screening visit;
   3. Fibrous changes in the lungs characteristic for COVID-19 confirmed by the chest CT scan at screening visit.
4. Negative COVID-19 screening test (confirmed).
5. Severity grade 2 (moderate) or 3 (severe) according to the mMRC Dyspnea Scale at the screening and randomization visits.
6. Decreased lung function FVC and/or DLCO <80% of the predicted value at the screening visit.
7. The patient's consent to use adequate contraception methods during the entire study and within 3 months after its completion. The adequate contraception methods include the use of the following:

   * oral or transdermal contraceptives;
   * condom or diaphragm (barrier method) with spermicide;
   * intrauterine device.

Exclusion Criteria:

1. Pregnant or breastfeeding women, or women planning pregnancy during the clinical study; women with childbearing potential (including those who have not been sterilized by surgery and in the postmenopausal period for less than 2 years) who do not use adequate contraception methods.
2. The use of invasive artificial lung ventilation (iALV), plasma transfusion (including plasma of convalescents) and other blood components during therapy against COVID-19.
3. Chronic airway disease in the past medical history, including idiopathic pulmonary fibrosis (IPF), bronchial asthma, chronic obstructive pulmonary disease (COPD), or pulmonary hypertension, diagnosed before COVID-19.
4. Significant cardiovascular diseases at present time or during 6 months prior to the screening, including: chronic heart failure class III or IV (according to the New York Heart Association classification), clinically significant ventricular arrhythmias (ventricular tachycardia, ventricular fibrillation), unstable angina, myocardial infarction, heart and coronary surgery, significant heart valves disease, uncontrolled hypertension with systolic blood pressure> 180 mm Hg and diastolic blood pressure> 110 mm Hg, thromboembolia of the pulmonary artery or deep vein thrombosis
5. Nephrotic syndrome, moderate to severe chronic renal failure, or significant kidney disease with a glomerular filtration rate (GFR) <60 ml/min at the screening visit.
6. Cirrhosis of the liver in the past medical history; increase in alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) by 3 or more times from the upper normal level (UNL) at the screening visit; an increase in the total bilirubin level by 2 or more times from UNL at the screening visit.
7. Hemoglobin level <90 g/L at the screening visit.
8. Severe diseases of the central nervous system, including seizures or conditions in the past medical history that can cause their development; stroke or transient ischemic attack within 6 months prior to the screening visit; traumatic brain injury or loss of consciousness within 6 months prior to the screening visit; a brain tumor.
9. Signs of severe uncontrolled intercurrent disease, such as disorders of the nervous system, kidney, liver, endocrine system and gastrointestinal tract, which, in the opinion of the Investigator, could interfere with the patient's participation in the study.
10. Malignant neoplasms requiring chemotherapy treatment within 6 months prior to the screening visit.
11. HIV infection in the past-medical history.
12. Prostate cancer or benign prostatic hyperplasia (BPH) with residual urine volume of more than 100 ml in the past medical history of men.
13. Hypersensitivity or intolerance to any component of the investigated drug.
14. Participation in other clinical studies within 2 months prior to the screening visit.
15. Administration of the following medications: bronchodilators, anticholinergics, corticosteroids, cytostatics, colchicine, cyclosporin A, interferon-γ-1b, bosentan, macitentan, etanercept, sildenafil, imatinib, n-acetylcysteine, warfarin, ambrisentan, nintedanib, pirfenidone 1 month prior to the screening visit.
16. Inability to read or write; unwillingness to understand and follow the procedures of the study protocol; noncompliance with the drugs administration or procedures schedule, which according to the researchers may affect the study results or the patient safety and prevent the further participation of the patient in the study; any other associated medical or serious mental conditions that make the patient inadequate for participation in the clinical study and restrict the validity of informed consent or may affect the patient's ability to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-10 (Actual)

PRIMARY OUTCOMES:
Rate of clinically significant change in FVC and/or DLCO at Week 4 relative to the baseline value | Day 1- Day 28
  Clinically significant changes include a relative ≥ 10% increase in FVC or a relative increase in FVC within the range from ≥ 5% to <10% and a relative ≥ 15% in DLCO

SECONDARY OUTCOMES:
Change in distance covered for 6 minutes (6MWD) at Weeks 2 and 4 from the baseline value (based on 6-minute walk test) | Day 1- Day 28
Change in the score of the Borg scale at Weeks 2 and 4 from the baseline value (based on the 6-minute walk test) | Day 1- Day 28
Change in forced expiratory volume for the first second (FEV1) according to spirometry data at Weeks 1, 2, 3 and 4 relative to the baseline values | Day 1- Day 28
Change in FVC according to spirometry data at Weeks 1, 2, 3 and 4 relative to the baseline values | Day 1- Day 28
Change in FEV1/FVC according to spirometry data at Weeks 1, 2, 3 and 4 relative to the baseline values | Day 1- Day 28
Change in DLCO according to bodyplethysmography at Week 2 and Week 4 relative to baseline values | Day 1- Day 28
Change in Total Lung Capacity (TLC) according to bodyplethysmography at Week 2 and Week 4 relative to baseline values | Day 1- Day 28
Change in Functional Residual Capacity (FRC) according to bodyplethysmography at Week 2 and Week 4 relative to baseline values | Day 1- Day 28
The rate of reduction in the lung damage degree based on the computed tomography (CT) at Week 4 relative to the baseline value | Day 1- Day 28
  Classification of lung damage includes the following stages: CT-0 (norm), CT-1 (< 25% of lung damage), CT-2 (25-50% of lung damage), CT-3 (50-75% of lung damage), CT-4 (> 75% of lung damage)
Change in mMRC Dyspnea Score in Week 1, Week 2, Week 3, and Week 4 from the baseline value | Day 1- Day 28
Change in the overall score of the KBILD Questionnaire at Week 2 and Week 4 relative to the baseline value | Day 1- Day 28

OTHER OUTCOMES:
The rate of adverse events (AEs) | Day 1- Day 28
The rate of serious adverse events (SAEs) | Day 1- Day 28
Residual concentration Ctrough of the active substance of Treamid | Day 1- Day 28
  Blood sampling for the PK study of the parameter Сtrough will be performed for all patients prior to administration of the Treamid / Placebo at Week 0, Week 2, and Week 4 visits.

CONTACTS AND LOCATIONS:
Locations (8):
- Russia (8):
  - Federal State-Funded Research Institution "Research Institute of Complex Cardiovascular Diseases", Kemerovo
  - Federal State Budgetary Institution "N.N. Burdenko Military Clinical Hospital", Moscow
  - SBEI HPE The First Moscow State Medical University n.a. Sechenov of Ministry of Health of Russian Federation, University Hospital #2, Department of Development of New Medicines, Moscow
  - Moscow State Medical-Dentist University n.a. A.I. Evdokimov on basis of SMHI "City Hospital № 62", branch 5, Moscow
  - State Budgetary Health Institution "Republican Hospital named V.A.Baranov", Petrozavodsk
  - Federal State Budgetary Educational Institution of Higher Education "Rostov State Medical University", Rostov-on-Don
  - LLC "Medical Center "Reavita Med St. Petersburg", Saint Petersburg
  - State autonomous healthcare institution of Yaroslavl Region "Сlinical hospital for emergency medical care n. a. N.V. Solovyov", Yaroslavl

REFERENCES:
- [Derived] Bazdyrev E, Panova M, Brachs M, Smolyarchuk E, Tsygankova D, Gofman L, Abdyusheva Y, Novikov F. Efficacy and safety of Treamid in the rehabilitation of patients after COVID-19 pneumonia: a phase 2, randomized, double-blind, placebo-controlled trial. J Transl Med. 2022 Nov 3;20(1):506. doi: 10.1186/s12967-022-03660-9. PMID 36329513